CLINICAL TRIAL: NCT02025257
Title: Effects of Exercise in Patients With Coronary Artery Disease Aged 80 Years or Older - a Randomized Controlled Trial
Brief Title: Effects of Exercise in Patients With Coronary Artery Disease Aged 80 Years or Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Bäck, Phd, RPT, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 462-13
Record Dates: First submitted 2013-10-21; First posted 2014-01-01 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; elderly; exercise; exercise-based cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Individually prescribed hospital based exercise in group two times a week, home-based exercise once a week. The exercise intervention consists of interval based aerobic exercise on a bicycle ergometer 30 minutes with intensity level at 13-17 at Borg scale, resistance exercises and balance exercises
  Interventions: Other: Exercise
- Control (No Intervention): Patients are asked to live as usual.

INTERVENTIONS:
Other: Exercise — Individually prescribed hospital based exercise in group two times a week, home-based exercise once a week. The exercise intervention consists of interval based aerobic exercise on a bicycle ergometer 30 minutes with intensity level at 13-17 at Borg scale, resistance exercises and balance exercises
  Arms: Exercise

SUMMARY:
The purpose of this study is to investigate the effects of exercise for patients with coronary artery disease (CAD) aged 80 years and older, with special reference to maximum aerobic capacity, muscle endurance, physical functioning, level of physical activity, health related quality of life, anxiety, depression and endothelial function, compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute coronary artery disease
* Aged 80 years or older

Exclusion Criteria:

* Inability to understand or speak the Swedish language
* Serious physical or psychological disease interfering with participation in an exercise intervention
* Patients are already exercising three times or more/week

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-12; Primary Completion 2019-05 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Change in maximum aerobic capacity | At baseline and after 4 months
  A maximum exercise test on an electronically braked cycle ergometer, with watts as marker of maximum aerobic capacity.

SECONDARY OUTCOMES:
Change in level of physical activity | At baseline and after 4 months
  Level of physical activity will be measured by an accelerometer and an activity diary
Change in muscular endurance | At baseline and after 4 months
  Will be measured by three clinical endurance tests including unilateral isotonic heel lift, unilateral isotonic shoulder flexion, bilateral isometric shoulder abduction
Change in physical functioning | At baseline and after 4 months
  Including tests of balance: short physical performance battery, one leg standing, timed up and go, and the activities specific balance confidence scale.
Change in health related quality of life | At baselline and after 4 months
  measured by a self-rated health questionnaire
Change in anxiety and depression | At baseline and after 4 months
  measured by the hospital anxiety and depression scale
Change in endothelial function | At baseline and after 4 months
  Evaluated with non-invasive ultrasound
Change in transthoracic evaluation of resting coronary flow velocity | At baseline and after 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bäck, PhD, Principal Investigator — Department of Physiotherapy, Sahlgrenska University Hospital, Gothenburg, Sweden; Per Albertsson, PhD, Study Chair — Department of Cardiology, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Department of physiotherapy, Sahlgrenska University Hospital, Gothenburg, Select A State…, Sweden

REFERENCES:
- [Result] Brosved M, Hirlekar G, Philip Wigh J, Sundberg H, Ziden L, Karlsson T, Albertsson P, Back M. Effects of Cardiac Rehabilitation on Physical Fitness, Physical Function, and Self-reported Outcomes in Patients >/=80 yr: A RANDOMIZED CONTROLLED TRIAL. J Cardiopulm Rehabil Prev. 2022 Sep 1;42(5):331-337. doi: 10.1097/HCR.0000000000000683. Epub 2022 Mar 31. PMID 35362694